CLINICAL TRIAL: NCT03054129
Title: Efficacy of Balance Training in Patients With Rotator Cuff Disease: A Randomized Controlled Trial
Brief Title: Efficacy of Balance Training in Patients With Rotator Cuff Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ertan Sahinoglu, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2110-GOA
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Results first posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-03

CONDITIONS: Rotator Cuff Injury
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation and balance training (Experimental): Each patient will attend rehabilitation program for three days per week for six weeks. Patients will receive balance training in addition to supervised rehabilitation program which is including patient education, stretching and strengthening exercises.
  Patients will also implement home exercise program. Balance training will be non-supervised program.
  Interventions: Other: Rehabilitation and balance training
- Rehabilitation program (Active Comparator): Each patient will attend rehabilitation program for three days per week for six weeks.
  Patients will receive supervised rehabilitation program which is including patient education, stretching and strengthening exercises.
  Patients will also implement home exercise program.
  Interventions: Other: Rehabilitation program

INTERVENTIONS:
Other: Rehabilitation and balance training — Stretching will be applied as hold-relax technique in Proprioceptive Neuromuscular Facilitation for shoulder flexion, abduction, internal and external rotations. Isotonic exercises will be done with elastic bands for strengthening.
  Home exercises will include postural, stretching and strengthening exercises. Balance exercises will receive as non-supervised program.
  Arms: Rehabilitation and balance training
Other: Rehabilitation program — Rehabilitation program will be same in this group except balance exercises.
  Arms: Rehabilitation program

SUMMARY:
The purpose of the study is to determine whether balance training is effective in patients with rotator cuff disease.

ELIGIBILITY:
Inclusion Criteria:

* Verification of the diagnosis of rotator cuff disease by a medical practitioner via radiological techniques.
* Pain due to unilateral rotator cuff disease at least four weeks.

Exclusion Criteria:

* Systemic pathology including inflammatory joint disease.
* More than %50 restriction of passive range of motion in two or more planes.
* History of major surgery on the lower extremities and shoulder regions.
* Acute or chronic pain in the spine or lower extremities.
* An injury of the lower extremities during the last six months which affected functional capabilities.
* Any kind of neurological complaint.
* Cardiovascular diseases which affect balance.
* Acute dizziness
* Medications which affected balance
* Subjects who performed balance training

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ertan ŞAHİNOĞLU, MSc, Principal Investigator — Dr. İsmail Atabek Physical Therapy and Rehabilitation Center; Bayram ÜNVER, PhD, Study Director — Dokuz Eylul University, School of Physical Therapy and Rehabilitation; Serkan ERKUŞ, MD, Principal Investigator — Tepecik Training and Research Hospital; Kamil Yamak, MD, Principal Investigator — University of Health Sciences, İzmir Bozyaka Education and Research Hospital
Locations (1):
- Dr. İsmail Atabek Physical Therapy and Rehabilitation Center, Izmir, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Groups:
- Rehabilitation Program: Each patient will attend rehabilitation program for three days per week for six weeks.
  Patients will receive supervised rehabilitation program which is including patient education, stretching and strengthening exercises.
  Patients will also implement home exercise program.
  Rehabilitation program: Rehabilitation program will be same in this group except balance exercises.
- Rehabilitation and Balance Training: Each patient will attend rehabilitation program for three days per week for six weeks. Patients will receive balance training in addition to supervised rehabilitation program which is including patient education, stretching and strengthening exercises.
  Patients will also implement home exercise program. Balance training will be non-supervised program.
  Rehabilitation and balance training: Stretching will be applied as hold-relax technique in Proprioceptive Neuromuscular Facilitation for shoulder flexion, abduction, internal and external rotations. Isotonic exercises will be done with elastic bands for strengthening.
  Home exercises will include postural, stretching and strengthening exercises. Balance exercises will receive as non-supervised program.
Period: Overall Study
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Started | 21 | 21
Completed | 19 | 20
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46 [42.5 to 51.5] | 50 [42 to 56.25] | 49 [42.5 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 16
  Male | 14 | 9 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 27.54 [23.68 to 28.22] | 25.90 [24.77 to 28.96] | 25.95 [24.09 to 28.50]
Employment status [Number; unit: participants]
  Working | 15 | 11 | 26
  Not working | 0 | 6 | 6
  Retired | 4 | 3 | 7
Education level [Number; unit: participants]
  Less than high school | 8 | 4 | 12
  High school graduate | 5 | 6 | 11
  College graduate | 6 | 10 | 16
Smoking habit [Number; unit: participants]
  Smoker | 10 | 11 | 21
  Nonsmoker | 9 | 9 | 18
Affected shoulder [Number; unit: participants]
  Dominant | 15 | 11 | 26
  Nondominant | 4 | 9 | 13
Comorbidities [Number; unit: participants]
  Hypertension | 0 | 5 | 5
  Diabetes mellitus | 1 | 2 | 3
  Lung disease | 0 | 1 | 1
  Other medical problems | 0 | 3 | 3
  No comorbidity | 18 | 9 | 27
Diagnosis [Number; unit: participants]
  Supraspinatus full thickness tear | 3 | 1 | 4
  Supraspinatus partial thickness tear | 7 | 8 | 15
  Supraspinatus+infraspinatus partial thickness tear | 2 | 0 | 2
  Supraspinatus tendinopathy | 1 | 2 | 3
  Supraspinatus + subscapularis tendinopathy | 0 | 1 | 1
  Subacromial impingement syndrome | 6 | 8 | 14
Pain duration [Median (Inter-Quartile Range); unit: weeks] | 16 [14 to 26] | 22 [9.50 to 36] | 20 [12 to 30]

OUTCOME MEASURES:

1. Primary Outcome: Postural Control-Stability Index in Solid Surface - Eyes Open
Description: Stability Index obtained by Tetrax Interactive Balance System No specified a minimum and maximum value. A lower score indicates better postural stability.
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: In rehabilitation program group, two patients withdrew from study In rehabilitation and balance training group, one patients excluded from the study due to a sytemic disease diagnosed.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale | 1.06 [-0.74 to 3] | 2.00 [-1.99 to 3.36]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.866, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Postural Control-Stability Index in Solid Surface - Eyes Closed
Description: as for outcome 1
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale | 0.74 [-2.96 to 3.53] | -2.37 [-5.35 to 3.00]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.361, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change of Quality of Life
Description: Change of Western Ontario Rotator Cuff Index score Total score range 0 (worst) to 2,100 (best).
Time Frame: Before treatment and 6 weeks (end treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale | 42.38 [21.43 to 52.86] | 36.43 [23.69 to 48.21]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.565, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Functional Limitations
Description: Change of Shoulder Pain and Disability Index score Total score 0-100. A higher score indicates worse pain and disability.
Time Frame: Before treatment and 6 weeks (end treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale
  Before treatment-Pain | 70.00 [52.00 to 82.00] | 76.00 [64.00 to 82.00]
  Before treatment-Disability | 47.50 [26.25 to 60.62] | 53.75 [38.12 to 73.12]
  Before treatment-Total | 60.00 [35.76 to 70.00] | 64.58 [49.22 to 78.28]
  After treatment-Pain | 4.00 [1.00 to 26.00] | 17.00 [8.00 to 40.00]
  After treatment-Disability | 2.50 [0.00 to 10.00] | 10.00 [2.50 to 25.62]
  After treatment-Total | 5.38 [1.15 to 16.54] | 15.38 [4.42 to 32.08]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Other; p = 0.000, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change of Pain
Description: Change of numeric rating scale score (activity, rest and night) 0 = no pain, 10 = worst possible pain
Time Frame: Before treatment and 6 weeks (end treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
units on a scale
  Before treatment-on movement | 5 [4 to 6] | 7 [5.75 to 8]
  Before treatment-at rest | 0 [0 to 3] | 0.50 [0 to 4]
  Before treatment-at night | 6 [5 to 8] | 7 [5 to 8]
  After treatment-on movement | 0 [0 to 1] | 1 [0 to 2.25]
  After treatment-at rest | 0 [0 to 0] | 0 [0 to 0]
  After treatment-at night | 0 [0 to 0.50] | 0.50 [0 to 2]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Other; p = 0.000, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Cognitive State
Description: Cognitive functioning of patients assessed by Mini Mental State Examination Score range 0 (worst) to 30 (best).
Time Frame: Only before treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale | 25 [24 to 27.5] | 26 [24 to 29]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.357, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Postural Control-Stability Index in Standing on Pillows - Eyes Open
Description: as for outcome 1
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale | 1.40 [-2.66 to 3.15] | 0.71 [-1.27 to 4.50]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.715, Wilcoxon (Mann-Whitney)

8. Primary Outcome: Postural Control-Stability Index in Standing on Pillows - Eyes Closed
Description: as for outcome 1
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale | -0.52 [-3.85 to 2.02] | -0.31 [-8.55 to 8.02]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.978, Wilcoxon (Mann-Whitney)

9. Primary Outcome: Postural Control-Stability Index in Head Turned Right 45° - Eyes Closed
Description: as for outcome 1
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale | 2.42 [0.27 to 3.48] | 0.61 [-3.49 to 3.38]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.191, Wilcoxon (Mann-Whitney)

10. Primary Outcome: Postural Control-Stability Index in Head Turn Left About 45° - Eyes Closed
Description: as for outcome 1
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale | 2.62 [0.15 to 4.35] | -0.33 [-4.31 to 2.89]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.097, Wilcoxon (Mann-Whitney)

11. Primary Outcome: Postural Control-Stability Index in Head Raised Backward 30° - Eyes Closed
Description: as for outcome 1
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale | 2.15 [-0.86 to 4.65] | 2.42 [-4.83 to 4.81]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.339, Wilcoxon (Mann-Whitney)

12. Primary Outcome: Postural Control-Stability Index in Head Downward 30° - Eyes Closed
Description: as for outcome 1
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale | 1.88 [0.25 to 4.48] | -0.48 [-3.96 to 2.15]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.016, Wilcoxon (Mann-Whitney)

13. Primary Outcome: Postural Control-Fourier Transformation (F5) in Solid Surface - Eyes Open
Description: Fourier transformation obtained by Tetrax Interactive Balance System No specified a minimum and maximum value. A lower value indicates higher stability
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hz
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
Hz | 0.29 [-0.53 to 0.90] | 0.16 [-0.13 to 0.73]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.933, Wilcoxon (Mann-Whitney)

14. Primary Outcome: Postural Control-Fourier Transformation (F5) in Solid Surface - Eyes Closed
Description: as for outcome 13
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hz
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
Hz | 0.04 [-0.33 to 0.58] | -0.72 [-1.39 to 0.70]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.136, Wilcoxon (Mann-Whitney)

15. Primary Outcome: Postural Control-Fourier Transformation (F5) in Standing on Pillows - Eyes Open
Description: as for outcome 13
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hz
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
Hz | -0.55 [-0.71 to 1.29] | 0.07 [-0.57 to 0.67]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.673, Wilcoxon (Mann-Whitney)

16. Primary Outcome: Postural Control-Fourier Transformation (F5) in Standing on Pillows - Eyes Closed
Description: as for outcome 13
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hz
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
Hz | -0.67 [-1.30 to 0.09] | -1.03 [-3.20 to 1.73]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.715, Wilcoxon (Mann-Whitney)

17. Primary Outcome: Postural Control-Fourier Transformation (F5) in Head Turned Right 45° - Eyes Closed
Description: as for outcome 13
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hz
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
Hz | 1.04 [-0.08 to 1.87] | -0.35 [-1.50 to 0.69]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.040, Wilcoxon (Mann-Whitney)

18. Primary Outcome: Postural Control-Fourier Transformation (F5) in Head Turn Left About 45° - Eyes Closed
Description: as for outcome 13
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hz
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
Hz | 0.19 [-0.30 to 0.87] | 0.25 [-0.50 to 1.48]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.779, Wilcoxon (Mann-Whitney)

19. Primary Outcome: Postural Control-Fourier Transformation (F5) in Head Raised Backward 30° - Eyes Closed
Description: as for outcome 13
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hz
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
Hz | 0.63 [0.16 to 1.29] | -0.21 [-0.98 to 1.01]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.152, Wilcoxon (Mann-Whitney)

20. Primary Outcome: Postural Control-Fourier Transformation (F5) in Head Downward 30° - Eyes Closed
Description: as for outcome 13
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hz
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
Hz | 0.07 [-0.46 to 0.97] | -0.54 [-1.74 to 0.60]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.129, Wilcoxon (Mann-Whitney)

21. Primary Outcome: Postural Control-Fourier Transformation (F6) in Solid Surface - Eyes Open
Description: as for outcome 13
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hz
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
Hz | 0.24 [-0.10 to 0.74] | 0.14 [-0.38 to 0.45]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.384, Wilcoxon (Mann-Whitney)

22. Primary Outcome: Postural Control-Fourier Transformation (F6) in Solid Surface - Eyes Closed
Description: as for outcome 13
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hz
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
Hz | 0.04 [-0.54 to 0.97] | 0.22 [-0.86 to 1.13]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.978, Wilcoxon (Mann-Whitney)

23. Primary Outcome: Postural Control-Fourier Transformation (F6) in Standing on Pillows - Eyes Open
Description: as for outcome 13
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hz
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
Hz | -0.12 [-0.66 to 0.88] | 0.27 [-0.75 to 1.14]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.715, Wilcoxon (Mann-Whitney)

24. Primary Outcome: Postural Control-Fourier Transformation (F6) in Standing on Pillows - Eyes Closed
Description: as for outcome 13
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hz
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
Hz | -0.42 [-1.21 to 0.77] | 0.83 [-2.04 to 1.68]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.546, Wilcoxon (Mann-Whitney)

25. Primary Outcome: Postural Control-Fourier Transformation (F6) in Head Turned Right 45° - Eyes Closed
Description: as for outcome 13
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hz
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
Hz | -0.02 [-0.36 to 0.60] | 0.14 [-0.97 to 1.09]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.933, Wilcoxon (Mann-Whitney)

26. Primary Outcome: Postural Control-Fourier Transformation (F6) in Head Turn Left About 45° - Eyes Closed
Description: as for outcome 13
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hz
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
Hz | 0.04 [-0.44 to 0.52] | 0.04 [-0.77 to 0.66]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.684, Wilcoxon (Mann-Whitney)

27. Primary Outcome: Postural Control-Fourier Transformation (F6) in Head Raised Backward 30° - Eyes Closed
Description: as for outcome 13
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hz
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
Hz | 0.18 [-0.06 to 1.03] | -0.23 [-0.84 to 0.43]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.112, Wilcoxon (Mann-Whitney)

28. Primary Outcome: Postural Control-Fourier Transformation (F6) in Head Downward 30° - Eyes Closed
Description: as for outcome 13
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hz
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
Hz | 0.44 [-0.18 to 1.20] | -0.25 [-1.28 to 0.43]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.012, Wilcoxon (Mann-Whitney)

29. Primary Outcome: Postural Control-Weight Distribution Index in Solid Surface - Eyes Open
Description: Weight Distribution Index obtained by Tetrax Interactive Balance System No specified a minimum and maximum value. A lower value indicates higher stability.
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale | -0.43 [-2.13 to 1.41] | 0.47 [-2.43 to 2.16]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.633, Wilcoxon (Mann-Whitney)

30. Primary Outcome: Postural Control-Weight Distribution Index in Solid Surface - Eyes Closed
Description: as for outcome 29
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale | 0.11 [-1.32 to 1.74] | -0.62 [-1.61 to 1.03]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.736, Wilcoxon (Mann-Whitney)

31. Primary Outcome: Postural Control-Weight Distribution Index in Standing on Pillows - Eyes Open
Description: as for outcome 29
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale | -1.74 [-2.81 to 0.36] | -0.19 [-2.53 to 2.64]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.227, Wilcoxon (Mann-Whitney)

32. Primary Outcome: Postural Control-Weight Distribution Index in Standing on Pillows - Eyes Closed
Description: as for outcome 29
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale | -1.57 [-2.39 to 0.01] | 1.21 [-1.81 to 4.39]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.109, Wilcoxon (Mann-Whitney)

33. Primary Outcome: Postural Control-Weight Distribution Index in Head Turned Right 45° - Eyes Closed
Description: as for outcome 29
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale | -0.25 [-2.37 to 1.39] | -0.35 [-0.91 to 0.35]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.844, Wilcoxon (Mann-Whitney)

34. Primary Outcome: Postural Control-Weight Distribution Index in Head Turn Left About 45° - Eyes Closed
Description: as for outcome 29
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale | -1.97 [-2.91 to -0.67] | -0.57 [-1.72 to 0.27]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.122, Wilcoxon (Mann-Whitney)

35. Primary Outcome: Postural Control-Weight Distribution Index in Head Raised Backward 30° - Eyes Closed
Description: as for outcome 29
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale | -0.71 [-2.19 to 1.75] | -0.91 [-3.26 to 1.86]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.715, Wilcoxon (Mann-Whitney)

36. Primary Outcome: Postural Control-Weight Distribution Index in Head Downward 30° - Eyes Closed
Description: as for outcome 29
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale | -0.47 [-2.52 to 0.39] | -0.81 [-1.74 to 2.44]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.593, Wilcoxon (Mann-Whitney)

37. Primary Outcome: Postural Control-Fall Index
Description: Fall Index obtained by Tetrax Interactive Balance System Minimum value = 0, Maximum value = 100. A higher value indicating a greater chance of falling.
Time Frame: Before treatment and 6 weeks (end of the treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
Number analyzed (Participants) | 19 | 20
score on a scale | -2.00 [-10.00 to 12.00] | -1.00 [-10.50 to 10.50]
Statistical Analysis 1: Comparison: Rehabilitation Program vs Rehabilitation and Balance Training; Test type: Superiority; p = 0.508, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: No adverse effects were expected in the study; therefore, it adverse events were not collected.
Description: No adverse effects were expected in the study.; therefore, it adverse events were not collected.
Arm/Group | Rehabilitation Program | Rehabilitation and Balance Training
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/29/NCT03054129/Prot_SAP_000.pdf